CLINICAL TRIAL: NCT03044145
Title: The Cultural Formulation Interview-Engagement Aid for Mental Health Treatment
Brief Title: The Cultural Formulation Interview-Engagement Aid
Acronym: CFI-EA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Neil Krishan Aggarwal, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 7234; 1K23MH102334 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Communication; Adherence, Patient
Keywords: Cultural Competence; Patient-Clinician communication
MeSH Terms: conditions — Communication; Patient Compliance | interventions — Reoperation; Therapeutics

STUDY DESIGN:
Intervention Model Description: This study follows an NIMH model known as the Stage Model of Intervention Development. The first project is creating a cross-cultural communication intervention designed to improve patient adherence in mental health services through patient and clinician feedback at JHMC and expert consensus with my K23 mentoring team. The second project is testing the intervention in a trial that compares the CFI-EA to treatment as usual.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Project 1: The Cultural Formulation Interview-Engagement Aid (Experimental): The first project is creating the intervention through patient and clinician feedback at JHMC and expert consensus with the K23 mentoring team. The CFI-EA is a list of questions that clinicians can use to customize patient treatment plans based on a cultural competence assessment.
  Interventions: Behavioral: The Cultural Formulation Interview-Engagement Aid
- Project 2: The Cultural Formulation Interview-Engagement Aid (Experimental): In this arm the study team will test the revised CFI-EA against treatment as usual in a pilot trial.
  Interventions: Behavioral: The Cultural Formulation Interview-Engagement Aid (Revised)
- Project 2: Treatment as usual (Active Comparator): Treatment as usual at JHMC consists of clinicians creating treatment plans for patients without any specific training in medical communication or treatment negotiation.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: The Cultural Formulation Interview-Engagement Aid — Culture affects how all people communicate and understand the world. Culture is important because patients and clinicians from different cultural backgrounds may have different preferences for communication. Mismatch in the clinician's approach and the patient's expectations of care can lead to patient dissatisfaction and discontinuation with treatment. Patients and clinicians may also have different views about what caused an illness, how it functions, what makes it better or worse, and the types of treatment needed. The CFI-EA is a series of questions over three sessions that clinicians can use to clarify patient views about treatment and communication so that patients stay in treatment longer. Clinicians can use the CFI-EA to customize their current treatment plans.
  Arms: Project 1: The Cultural Formulation Interview-Engagement Aid
Behavioral: The Cultural Formulation Interview-Engagement Aid (Revised) — The study team will revise the CFI-EA based on patient and clinician feedback. The study team expects that the revisions will consist of changes to the questions such as adding or subtracting specific items or revising the wording of the content. The study team do not anticipate other changes, though we will let our empirical data analyses guide revisions in consultation with the K23 mentor team.
  Arms: Project 2: The Cultural Formulation Interview-Engagement Aid
Behavioral: Treatment as usual — Standard mental health treatment at FHMC
  Arms: Project 2: Treatment as usual

SUMMARY:
This study consists of two projects:

Project 1: The study team will create and refine the CFI-EA by enrolling 3 clinicians and 9-12 patients to test the CFI-EA's feasibility and acceptability from patient and clinician feedback in a pre-pilot trial. The study team will first train clinicians in the CFI-EA by reading over the CFI-EA treatment manual and practicing how they can use it in behavioral simulations, and then check whether participants think they can do it (feasibility) and like it (acceptability) through standard measures. Following this the study team will revise the CFI-EA based on their feedback for the comparative open trial in Phase 2.

Project 2: The study team will test the revised CFI-EA against treatment as usual in a pilot trial. 3 clinicians and 12-15 patients will be enrolled in each arm. As before, the study team will first train clinicians in the revised CFI-EA by reading over the CFI-EA treatment manual and practicing how they can use it in behavioral simulations. Then, the study team will check whether participants think they can do it (feasibility) and like it (acceptability) through standard measures, and in addition will also explore any initial effects on communication behaviors among patients and clinicians and treatment engagement based on treatment retention.

The specific aims are:

For Project 1:

1. To pretest the CFI-EA intervention in a mental health setting through a pre-pilot open trial that explores communication mechanisms of action in terms of communication behavior and cultural content, and
2. To revise the CFI-EA intervention based on patient and clinician feedback on its feasibility and acceptability.

As real-world community stakeholders for whom the CFI-EA is being developed, patients and clinicians can provide helpful perspectives on how the CFI-EA can help clinicians tailor treatment plans around patient cultural views and treatment preferences to keep patients in care. The CFI-EA will be revised around areas of maximal agreement among patients and clinicians with the help of health disparities and communication experts.

For Project 2:

1. To test the revised CFI-EA's feasibility and acceptability among patients and clinicians in a pilot open trial against treatment as usual, and
2. To explore the relationship between the revised CFI-EA's effects on patient-clinician communication and treatment engagement.

The study team hypothesize that clinicians using the revised CFI-EA will show more positive communication behaviors compared to clinicians delivering treatment as usual and that CFI-EA patients will stay in treatment longer. Communication behaviors will be assessed through communication analysis techniques such as the Roter Interaction Analysis System.

DETAILED DESCRIPTION:
Members of underserved racial/ethnic minority groups who participate more actively in the treatment process have almost three times the odds of staying in treatment and following up with appointments compared to standard treatment. Improving patient-clinician communication may therefore improve treatment engagement, from starting and participating in treatment actively to maintaining treatment for the successful resolution of symptoms and improvements in quality of life. Interventions that enhance communication behaviors by asking patients about their cultural views, using open-ended questions, establishing rapport, and using patient terms can increase patient participation and satisfaction. Interventions that expose clinicians to cultural content by asking patients about preferences for treatment, barriers to accessing services, the role of support from family or friends, and that encourage information exchange also improve treatment engagement. The goal of this study is to develop a communication intervention that improves treatment engagement for members of underserved racial and ethnic minority groups by improving clinician communication behaviors and exposing them to patient cultural content. Here, culture is understood as a dynamic process of meaning making between the patient and clinician. This intervention is not designed for patients belonging to a specific racial or ethnic group, but to improve general communication between patients and clinicians. The intervention improves communication by making communication behaviors and cultural content topics of explicit conversation rather than allowing clinicians to make cultural assumptions and take them for granted. We are focusing on racial and ethnic minorities because of significant evidence documenting disparities in health communication and care.

In session 1, the clinician does the full CFI in DSM-5 (~15 minutes) and then completes the full standard intake with information not already obtained through the CFI (~35 minutes). In sessions 2 and 3, the clinician integrates the CFI-EA (~5 minutes) within regular care in standard appointments. At JHMC, Session 2 lasts 60 minutes and is for treatment initiation. Session 3 lasts 20-30 minutes and is to check for treatment continuation. Because this is a grant to train in developing mental health interventions, the study team is following an NIMH model known as the Stage Model of Intervention Development. The first project is creating the intervention through patient and clinician feedback at JHMC and expert consensus with the K23 mentoring team. The second project is testing the intervention in a trial that compares the CFI-EA to treatment as usual. Patients for Project 1 will be recruited through a sample of convenience among patients accessing care on the days the research assistant is in the waiting area. For project 2, patients will be sampled consecutively by the JHMC's intake coordinator from the time that the project starts until the target enrollment is reached. The intake coordinator will keep a record of all patients who agree and do not agree to enroll in the study. Patients who agree to be enrolled during Project 2 will be recruited by the research assistant in the waiting area and then assigned randomly to either CFI-EA clinicians or treatment-as-usual clinicians based on a random number generator. The study team is using the same study measures in both projects to examine whether revisions to the CFI-EA conducted at the end of Project 1 show improvements in outcomes after Project 2.

ELIGIBILITY:
For Project 1

Inclusion Criteria:

* Male and female patients aged 18-80; Method of ascertainment: Self-report.
* New patients at JHMC, referred by the intake coordinator; Method of ascertainment: Intake coordinator.
* Willingness and ability to provide written informed consent after full explanation of study procedures. Method of ascertainment: RA informed consent interview that includes a capacity to consent screening form; Clinician referral.
* Racial and ethnic minority (African-American, Latino/Hispanic, Asian-American/Pacific Islander, and Native American). Method of ascertainment: Self-report

Exclusion Criteria:

* Actively suicidal or homicidal; Method of ascertainment: Self-report and clinician evaluation
* In need of acute detoxification services; Method of ascertainment: Self-report and clinician evaluation
* A condition that interferes with participation (i.e., dementia, mental retardation, or florid psychosis); Method of ascertainment: Clinician evaluation; patients ≥ 65 years of age will participate in a mini-cog exam.
* Caucasian race; Method of ascertainment: self-report

For Project 2

Inclusion Criteria:

* Male and female patients aged 18-80; Method of ascertainment: Self-report.
* New patients at JHMC, referred by the intake coordinator; Method of ascertainment: Intake coordinator.
* Willingness and ability to provide written informed consent after full explanation of study procedures. Method of ascertainment: RA informed consent interview that includes a capacity to consent screening form; Clinician referral.
* Racial and ethnic minority (African-American, Latino/Hispanic, Asian-American/Pacific Islander, and Native American). Method of ascertainment: Self-report

Exclusion Criteria:

* Actively suicidal or homicidal; Method of ascertainment: Self-report and clinician evaluation
* In need of acute detoxification services; Method of ascertainment: Self-report and clinician evaluation
* A condition that interferes with participation (i.e., dementia, mental retardation, or florid psychosis); Method of ascertainment: Clinician evaluation; patients ≥ 65 years of age will participate in a mini-cog exam.
* Caucasian race; Method of ascertainment: self-report
* Patients in Project 1 will be excluded from Participation in Project 2: Method of assessment: self-report and PI/RA evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
CFI-EA feasibility is defined as patient completion rates for all three sessions of the CFI-EA intervention. | two months after the third session
  CFI-EA feasibility is defined as patient completion rates for all three sessions of the CFI-EA intervention.
CFI-EA acceptability is defined as patient scores on the CSQ-8. | the third session
  CFI-EA acceptability is defined as patient scores on the CSQ-8.

SECONDARY OUTCOMES:
Treatment engagement defined as the percentage of patients staying within treatment 2 months after the third and last session of the CFI-EA has been delivered. | 2 months after the last session of the CFI-EA
  Defined as the percentage of patients staying within treatment 2 months after the third and last session of the CFI-EA has been delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Neil K Aggarwal, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Flushing Hospital Medical Center, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: No